CLINICAL TRIAL: NCT01672112
Title: Comparison of the Efficacy of Oral Oxycodone and Oral Codeine in the Treatment of Postcraniotomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Lim Pei-Pei Mandy, Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/02076
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Postcraniotomy Pain
Keywords: analgesic efficacy; oral codeine; oral oxycodone; postcraniotomy
MeSH Terms: interventions — Oxycodone; Codeine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Codeine (Other): Oral Codeine 60mg 6hrly/prn
  Interventions: Drug: Codeine
- Oxycodone (Active Comparator): Oral Oxycodone 5mg 6hrly/prn
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Oral Oxycodone 5mg 6hrly/prn
  Other Names: Oxynorm Immediate Release
  Arms: Oxycodone
Drug: Codeine — Oral Codeine 60mg 6hrly/prn
  Other Names: Codeine Phosphate
  Arms: Codeine

SUMMARY:
The efficacy of codeine is dependent on its demethylation to morphine. This extent of demethylation has wide inter-individual variability, making codeine's efficacy as a analgesic variable. Oxycodone is a semi-synthetic opioid and is a weak agonist on mu opioid receptors.

Codeine has been the mainstay of analgesia for patients after craniotomy for many years. Traditionally, craniotomies were not thought to be very painful procedures, hence the use of codeine, a moderately potent opioid (when compared to morphine).

However, in recent years, it has been found that up to 70% of post-craniotomy patients have moderate to severe pain and codeine did not provide adequate analgesic relief. Many studies have compared codeine to other drugs such as PCA morphine, fentanyl and tramadol, and patients on these stronger opioids generally had lower pain scores and better satisfaction.

No study has been conducted to determine the efficacy of analgesia of oral oxycodone to oral codeine.

Hence, the hypothesis is that oxycodone is more effective than codeine in providing pain relief in post-craniotomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-70 years of age
* Planned elective craniotomy
* ASA 1-3
* GCS 15 pre and post-op
* Able to understand and use the visual analogue scale

Exclusion Criteria:

* Patients with GCS < 15 pre and/or post-op.
* Patients who are unable to quantify pain according to VAS scale.
* Patients who will be left intubated post-op.
* Contraindications and/or allergies to any of the trial drugs.
* Patients with renal and/or hepatic impairment.
* Patients with decreased respiratory reserves.
* Patients with post-op cognitive dysfunction.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine the difference in the mean pain VAS scores in the oxycodone and codeine groups at 24hr. | 24hr post-op.

SECONDARY OUTCOMES:
To look at the incidence of adverse events in the oxycodone and codeine groups. | Up to 72hrs post-op.
  To compare the incidence of excessive sedation, respiratory depression and GCS; to compare the pain VAS scores at 48 and 72hrs post-op; to compare the mean satisfaction scores at 24 and 72hrs post-op.

CONTACTS AND LOCATIONS:
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore